CLINICAL TRIAL: NCT03684486
Title: Rehabilitation by Effort for Patients With Advanced Bronchial Cancer
Acronym: RehabKBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/11/0087
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Bronchial Cancer; Malignant Mesothelioma
Keywords: bronchial cancer; rehabilitation
MeSH Terms: conditions — Carcinoma, Bronchogenic; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rehabilitation by effort (Experimental): 8 sessions of rehabilitation by effort in sports medicine
  Interventions: Behavioral: rehabilitation by effort

INTERVENTIONS:
Behavioral: rehabilitation by effort

SUMMARY:
Bronchopulmonary cancers or mesothelioma are associated with effort deconditioning due to pathology (chronic inflammation) and also to treatments (surgery, radiotherapy, chemotherapy); it's considerably alters patients quality of life.

Investigators want to ensured the feasibility of rehabilitation by effort for these patients.

ELIGIBILITY:
Inclusion Criteria:

* General condition according to World Health Organisation 0-1
* Age between 18 and 70 years old
* Non progressive patients according to RECIST criteria 1.1 after chemotherapy treatment whichever line of treatment
* Autonomous patient
* Voluntary written informed consent signed
* Patients with social security insurance

Exclusion Criteria:

* Bone metastasis with fracture risk
* Significant cardiovascular pathology
* Cardiac, vascular, rheumatologic or neurologic contraindication
* Patients living far 60 kms from Toulouse
* Patients under juridical protection guardianship, or tutelage measure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
patients who completed at least 6 sessions of rehabilitation | 10 years
  number of patients who completed at least 6 sessions of rehabilitation by effort

CONTACTS AND LOCATIONS:
Overall Officials: Julien Mazières, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France